CLINICAL TRIAL: NCT04956497
Title: Registry Study of Extracorporeal Cardiopulmonary Resuscitation (eCPR) in China
Acronym: ECPR-China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-001
Record Dates: First submitted 2021-07-08; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-05

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Cardiopulmonary Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: extracorporeal membrane oxygenation (ECMO) — ECMO under ongoing cardiopulmonary resuscitation (eCPR) in patients with refractory cardiac arrest

SUMMARY:
The data of patients undergo extracorporeal cardiopulmonary resuscitation (eCPR) will be collected and analyzed. This study will provide useful information about the indication, the start time and others to improve the outcome of ECPR.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18y
* Cardiac arrested patients accept ECPR treatment

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (age>=18y) cardiac arrested patients accept ECPR treatment will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality rate | 28 days
  the death rate of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Jun Xu, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China